CLINICAL TRIAL: NCT01936623
Title: Computerized Brief Intervention vs. Delayed Computerized Brief Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01DA026003-B; 1R01DA026003 (NIH)
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-04

CONDITIONS: Drug Abuse
Keywords: brief intervention; computerized brief intervention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computerized Brief Intervention (Experimental): Computerized Brief Intervention is delivered using a talking, animated cartoon-like parrot that provides patient feedback, empathic reflection, and personalization regarding their drug use.
  Interventions: Behavioral: Computerized Brief Intervention
- Delayed Computerized Brief Intervention (Other): Participants receive only a substance abuse assessment at baseline. At three-month follow-up, they then receive the computerized brief intervention.
  Interventions: Behavioral: Computerized Brief Intervention

INTERVENTIONS:
Behavioral: Computerized Brief Intervention — No additional information needed.

SUMMARY:
The purpose of the study is to determine whether a computerized brief intervention for moderate risk drug use among adult primary care patients is more effective than providing such patients with a substance abuse assessment alone.

DETAILED DESCRIPTION:
The study will enroll 80 adult primary care patients who have moderate risk drug use. Eligible participants (N = 80) will be randomly assigned to immediately receive a computerized brief intervention focused on drug use or to receive the same computerized brief intervention at 3-month follow-up. All participants will be assessed at three time points: baseline, and at 3 and 6 month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* (1) minimum 18 years of age
* (2) primary care or dental patients at the participating clinics
* (3) score between 4 and 26 (moderate-risk) for illicit drug and/or nonmedical use of prescription drugs on any of the single item drug use risk scores of the ASSIST.

Exclusion Criteria:

* (1) score in the high-risk range on the ASSIST for any drug (except tobacco) or alcohol use (i.e., ASSIST score > 26)
* (2) no reported drug use within the past 3 months
* (3) drug abuse treatment within the past 12 months
* (4) a BI at the clinic with the behavioral health counselor within the past month
* (5) prior enrollment in the parent study;
* (6) plans to move out of New Mexico in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Schwartz, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- First Choice Community Healthcare, Edgewood, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Computerized Brief Intervention | Delayed Computerized Brief Intervention
Started | 40 | 40
Completed | 40 | 35
Not Completed | 0 | 5
Not completed — Lost to Follow-up | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Computerized Brief Intervention | Delayed Computerized Brief Intervention | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (12.4) | 36.0 (13.8) | 35.2 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 17 | 42
  Male | 15 | 23 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 19 | 34
  Not Hispanic or Latino | 25 | 21 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 33 | 36 | 69
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Alcohol, Smoking, and Substance Involvement Screening Tests (ASSIST) Global Continuum of Illicit Drug Risk Score
Description: The ASSIST Global Continuum of Illicit Drug Risk Score ranges from 0 to 308, with higher scores indicating greater risk.
Time Frame: 3 month follow-up
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Computerized Brief Intervention | Delayed Computerized Brief Intervention
Number analyzed (Participants) | 40 | 40
units on a scale | 24.4 (2.2) | 27.8 (2.2)

2. Secondary Outcome: Alcohol, Smoking, and Substance Involvement Screening Tests (ASSIST) Global Continuum of Illicit Drug Risk Score
Description: The ASSIST Global Continuum of Illicit Drug Risk Score ranges from 0 to 308, with higher scores indicating greater risk.
Time Frame: 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Computerized Brief Intervention | Delayed Computerized Brief Intervention
Number analyzed (Participants) | 40 | 40
units on a scale | 26.4 (2.2) | 27.1 (2.2)

3. Other Pre Specified Outcome: Number of Subjects Testing Positive on Hair Testing for Marijuana, Cocaine, Amphetamines, or Opioids.
Description: Radioimmunoassay (RIA) Tests were used.
Time Frame: 3-month
Population: Hair samples were missing due to refusal, insufficient quantity, and missing follow-up interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Computerized Brief Intervention | Delayed Computerized Brief Intervention
Number analyzed (Participants) | 19 | 16
Participants | 13 | 6

4. Other Pre Specified Outcome: Number of Subjects Positive on Hair Testing for Marijuana, Cocaine, Amphetamines, or Opioids
Description: Radioimmunoassay Testing (RIA) was conducted
Time Frame: 6-month follow-up
Population: Hair samples were missing due to refusal, insufficient quantity, and missing follow-up interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Computerized Brief Intervention | Delayed Computerized Brief Intervention
Number analyzed (Participants) | 21 | 14
Participants | 14 | 8

ADVERSE EVENTS:
Arm/Group | Computerized Brief Intervention | Delayed Computerized Brief Intervention
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes